CLINICAL TRIAL: NCT06560853
Title: Evaluation of a Comprehensive School Health Programme in Zambia: a Cluster-randomised Controlled Trial
Brief Title: Evaluation of a Comprehensive School Health Programme in Zambia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Economics and Political Science (Other)
Collaborators: University of Virginia (Other); Healthy Learners (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 264865
Record Dates: First submitted 2024-08-12; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Helminth Infection; Malaria; Schistosomiasis; Anemia; UTI; Diarrhea; Skin Rash; Cough
Keywords: School Health Services
MeSH Terms: conditions — Trematode Infections; Malaria; Schistosomiasis; Anemia; Diarrhea; Exanthema; Cough

STUDY DESIGN:
Intervention Model Description: Clusters (schools) are randomised to one of 3 treatment arms. Non-compliance with treatment or control is possible if participants move between schools. We expect low rates of transfers and will track any transfers which do occur.
Masking Description: Blinding of intervention units, i.e. schools, to their own treatment (or that of others) is not feasible. After the initial scoping and baseline data collection (during which treatment was masked to all participants and assessors), due to the nature of the intervention, there will be no blinding: both the beneficiaries and assessors monitoring the outcomes will be able to infer whether the school is receiving the HL programme or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- School health programme (SHP) (Experimental): SHP developed by Healthy Learners (HL) in collaboration with the Ministry of Education (MOE), which follows the WHO guidelines on school health activities. HL supports the upgrading of basic sanitation facilities and construction of a dedicated 'health room' in the school; trains selected teachers to become school health workers (SHWs) who deliver health and sanitation education, coordinate deworming and vitamin A supplementation in the school, and assess sick learners in the school health room using a clinical decision support system (CDSS), either treating in school or referring to the local health centre. At the health centre, children referred by SHWs are given priority by health care workers who see them within 30 minutes of arriving at the facility. Schools also create student networks (a "buddy" system) whereby learners monitor each other's absence and coordinate with SHWs, who can then follow up with the household.
  Interventions: Other: Comprehensive School Health Programme; Other: Deworming and vitamin A supplementation delivery
- Deworming and vitamin A supplementation (Active Comparator): Healthy Learners will enusre reliable delivery of the national deworming programme twice a year, during the same period as in the SHP arm, for comparability of the effect of prevention alone to the full SHP.
  Interventions: Other: Deworming and vitamin A supplementation delivery
- Status quo (No Intervention): Schools to operate as usual with no intervention other than the usual activities planned and organized by the government, as set out the 2006 School Health and Nutrition Policy, until the end of the trial.

INTERVENTIONS:
Other: Comprehensive School Health Programme — Combination intervention which consists of:
  * Upgrading sanitation facilities and constructing a 'health room' in the school
  * Health teacher training: 5-10 teachers per school are recruited and trained for two weeks to become School Health Workers (SHWs) by Healthy Learners
  * The SHWs: (1) deliver education on health and good sanitation and hygiene (2) coordinate with local clinics to deliver preventive care (e.g. school deworming and vitamin A supplementation); (3) assess sick students in the health room with a tablet-based clinical decision support system (CDSS); (4) treat sick students in the health room for some conditions (malaria, diarrhoea, schistosomiasis, pneumonia, conjunctivitis) or (5) refer to the health facility for treatment; (6) monitor absence of learners
  * Referral: learners referred by SHWs are given a referral form by the SHW, which contains information about symptoms and suggested diagnosis by the CDSS. The learners are prioritised in the local clinic.
  Other Names: SHP
  Arms: School health programme (SHP)
Other: Deworming and vitamin A supplementation delivery — Schools implement the government policy of distributing deworming drugs and vitamin A supplementation to learners twice a year. Additional support from Healthy Learners ensures reliable delivery.
  Other Names: Deworming
  Arms: Deworming and vitamin A supplementation; School health programme (SHP)

SUMMARY:
In Zambia, the health and well-being of children aged 5 to 14 has often been overlooked, leading to various health challenges affecting their development and education. The Healthy Learners (HL) program, in collaboration with the Zambian Government, aims to address this gap by implementing a comprehensive school health program. Trained teachers, known as school health workers (SHWs), play a key role by delivering health education, coordinating preventative care with local clinics, and overseeing a 'school health room' for sick students.

This study is a large cluster-randomized control trial in 225 schools. The goal of this trial is to compare the effects of the comprehensive school health programme (SHP) developed by HL against two alternatives: the current level of school health provision and the current school health activities enhanced with deworming and vitamin A coordination by HL, with their technical and financial support ensuring the reliable delivery of all health activities currently planned by the government.

1. What is the impact of the program on health-seeking, health, and education outcomes?
2. What are the indirect effects of the program on teachers and clinics?
3. What is the added value of such a comprehensive SHP, compared to (i) optimized (ii) or imperfect (status-quo) delivery of a limited range of school health activities (e.g., deworming and vitamin A supplements)?
4. How costly is the comprehensive SHP, and what factors affect its implementation?
5. What are the potential benefits of the program for long-term human capital accumulation (learning, well-being etc)?

ELIGIBILITY:
* Schools: eligible for SHP (not inaccessible in the rainy season, within 10km of health centre)
* School administrator: has at least one year experience in school and is the primary or deputy school manager (e.g., headteacher, deputy headteacher, senior teacher acting as financial officer)
* Learners: registered and in attendance in school during baseline, in grade 1, grade 3, or grade 5
* Parents, primary caregivers or guardians of selected learners. Guardians are eligible if they stay with the child and make schooling and health decisions for the child in the absence of parents/primary caregivers.
* Teachers: any teacher employed by study eligible schools (not volunteers)
* Health facilities: designated facilities in the catchment area of study schools
* Health facility staff: any staff doing OPD consultation present during facility data collection days

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28700 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Synthetic morbidity index | 18 months after intervention start
  Because the SHP delivers treatment of several diseases, we will create a composite disease burden index of the following outcomes:
  * malaria positive (using a rapid diagnostic test)
  * moderate to high worm load (using a stool test)
  * anaemia (using a hemocue test)
  * schistosomiasis (using a urine test)
  * diarrhoea in the past week (learner self-report) We test these outcomes in a randomly selected panel of 13,300 learners recruited at baseline, which ensures variety of age groups and balance of genders.
Average attendance rate over 24 months | 24 months after intervention start
  We will measure attendance during unannounced attendance spot checks (one per term over a 2-year period). Multiple measurements are required to capture seasonal variation. On each spot check visit, we will check attendance of a panel of learners randomly selected at baseline, which ensures variety of age groups and balance of genders. We will calculate each child's attendance rate across all the spot checks.

CONTACTS AND LOCATIONS:
Overall Officials: Mylene Lagarde, PhD, Principal Investigator — London School of Economics and Political Science; David Ross, PhD, Study Chair — University of Stellenbosch
Locations (6):
- Zambia (6):
  - Chingola District Education Board, Chingola, Copperbelt
  - Luanshya District Education Board, Luanshya, Copperbelt
  - Masaiti District Education Board, Masaiti, Copperbelt
  - Kawambwa District Education Board, Kawambwa, Luapula Province
  - Mwense District Education Board, Mwense, Luapula Province
  - Samfya District Education Board, Samfya, Luapula Province

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share a complete dataset at the individual-level containing all primary and secondary study outcomes, any other variables used in the analysis, and treatment assignments. Data will be anonymised to ensure no participants can be personally identified (directly or indirectly)
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available permanently. They will become available along with the publication of the study in a journal, as we will provide a replication package as part of the publication.

DOCUMENTS (2):
  • Study Protocol (2024-08-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT06560853/Prot_000.pdf
  • Informed Consent Form (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT06560853/ICF_001.pdf